CLINICAL TRIAL: NCT06413472
Title: Comparing Mechanical Power Values Using Geometric Methods at Different Inspiratory Rise and Pause Times: A Validation Study
Brief Title: Comparing Mechanical Power in Different Inspiratory Times
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other)
Responsible Party: Principal Investigator, Furkan Tontu, Doctor of Anesthesiology and Reanimation, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-Tslope
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Ventilator-Induced Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ARDS patients-PCV: Intubated patients with a diagnosis of ARDS in the intensive care unit, ventilated using Pressure-Controlled Ventilation (PCV).
  Interventions: Procedure: Mechanical ventilator adjustment for PCV
- ARDS patients-VCV: Intubated patients with a diagnosis of ARDS in the intensive care unit, ventilated using Volume-Controlled Ventilation (VCV).
  Interventions: Procedure: Mechanical ventilator adjustment for VCV

INTERVENTIONS:
Procedure: Mechanical ventilator adjustment for PCV — In pressure control ventilation (PCV) mode, patients will be ventilated for 5 minutes at a Tslope of 5% and another 5 minutes at 15% for both 1:1 and 1:2 I:E ratios. After each adjustment, screenshots of the mechanical ventilator (P-V loop screenshots) will be obtained . A total of 20 P-V loop screenshots will be captured over a 20-minute period (10 for the 1:2 ratio and 10 for the 1:1 ratio), which will be stored in the ventilators memory. The stored data will then be transferred from the ventilators memory to a computer via a flash drive.
  Groups: ARDS patients-PCV
Procedure: Mechanical ventilator adjustment for VCV — In volume control ventilation (VCV) mode, patients will be ventilated for 5 minutes at a Tslope of 5% and another 5 minutes at 15% for both 1:1 and 1:2 I:E ratios. After each adjustment, screenshots of the mechanical ventilator (P-V loop screenshots) will be obtained . A total of 20 P-V loop screenshots will be captured over a 20-minute period (10 for the 1:2 ratio and 10 for the 1:1 ratio), which will be stored in the ventilators memory. The stored data will then be transferred from the ventilators memory to a computer via a flash drive.
  Groups: ARDS patients-VCV

SUMMARY:
We aimed to compare mechanical power and energy values using geometric methods at varying inspiratory rise times.

DETAILED DESCRIPTION:
In this study, the researchers aim to compare the mechanical power and energy values calculated using the geometric method in Volume-Controlled Ventilation (VCV) and Pressure-Controlled Ventilation (PCV) modes at different inspiratory rise times.

ELIGIBILITY:
Inclusion Criteria:

* ARDS (Acute Respiratory Distress Syndrome) patients.
* Patients who are deeply sedated.
* Patients ventilated in:
* Pressure-Controlled Ventilation (PCV or PRVC) mode, or
* Volume-Controlled Ventilation (VCV) mode.
* Patients within the 24-48 hour period of their stay in the intensive care unit.

Exclusion Criteria:

* Patients with incomplete data.
* Patients diagnosed with:
* COPD (Chronic Obstructive Pulmonary Disease),
* Heart failure.
* Pregnant patients.
* Patients with a thoracopleural fistula.
* Hemodynamically unstable patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Patients with a diagnosis of ARDS in the general intensive care unit of the Anesthesiology and Reanimation Clinic at Bakırköy Dr. Sadi Konuk Training and Research Hospital."
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
MPgeo | 40 minute
  The mechanical power (MPgeo) values measured using the geometric method .
Energy | 40 minute
  Energy values measured using the geometric method .

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Background] Trinkle CA, Broaddus RN, Sturgill JL, Waters CM, Morris PE. Simple, accurate calculation of mechanical power in pressure controlled ventilation (PCV). Intensive Care Med Exp. 2022 May 30;10(1):22. doi: 10.1186/s40635-022-00448-5. PMID 35644896
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Background] Asar S, Acicbe O, Cukurova Z, Hergunsel GO, Canan E, Cakar N. Bedside dynamic calculation of mechanical power: A validation study. J Crit Care. 2020 Apr;56:167-170. doi: 10.1016/j.jcrc.2019.12.027. Epub 2020 Jan 2. PMID 31931417
- [Background] Giosa L, Busana M, Pasticci I, Bonifazi M, Macri MM, Romitti F, Vassalli F, Chiumello D, Quintel M, Marini JJ, Gattinoni L. Mechanical power at a glance: a simple surrogate for volume-controlled ventilation. Intensive Care Med Exp. 2019 Nov 27;7(1):61. doi: 10.1186/s40635-019-0276-8. PMID 31773328
- [Background] Chi Y, He H, Long Y. A simple method of mechanical power calculation: using mean airway pressure to replace plateau pressure. J Clin Monit Comput. 2021 Oct;35(5):1139-1147. doi: 10.1007/s10877-020-00575-y. Epub 2020 Aug 11. PMID 32780353
- [Background] Becher T, van der Staay M, Schadler D, Frerichs I, Weiler N. Calculation of mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Sep;45(9):1321-1323. doi: 10.1007/s00134-019-05636-8. Epub 2019 May 17. No abstract available. PMID 31101961
- [Background] van der Meijden S, Molenaar M, Somhorst P, Schoe A. Calculating mechanical power for pressure-controlled ventilation. Intensive Care Med. 2019 Oct;45(10):1495-1497. doi: 10.1007/s00134-019-05698-8. Epub 2019 Jul 29. No abstract available. PMID 31359082
- [Background] Asar S, Acicbe O, Sabaz MS, Kucur Tulubas E, Hergunsel GO, Cukurova Z, Canan E, Cakar N. Simplified calculation of mechanical power for pressure controlled ventilation in Covid-19 ARDS patients. Minerva Anestesiol. 2022 Jan-Feb;88(1-2):42-50. doi: 10.23736/S0375-9393.21.15741-4. PMID 35224956
- [Background] Acicbe O, Ozgur CY, Rahimi P, Canan E, Asar S, Cukurova Z. The effect of inspiratory rise time on mechanical power calculations in pressure control ventilation: dynamic approach. Intensive Care Med Exp. 2023 Dec 20;11(1):98. doi: 10.1186/s40635-023-00584-6. PMID 38117345
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452